CLINICAL TRIAL: NCT04702165
Title: Image - Navigated Resection of Lung Nodules
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Navigation Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2020P002692
Record Dates: First submitted 2020-12-23; First posted 2021-01-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Lung Diseases
Keywords: lung nodule; lung cancer; lung mass
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- VATS resection with J-bar (Experimental): Each patient with a lung nodule meeting criteria will undergo a lung resection which could be one of three approaches: iVATS with Dyna-CT, VATS, or open. Each approach will use a the experimental device the Lung Resection Marker Locator Kit
  Interventions: Device: lung resection with Lung Resection Marker Locator Kit

INTERVENTIONS:
Device: lung resection with Lung Resection Marker Locator Kit — Nodules eligible for surgical resection using the Lung Resection Marker Locator Kit

SUMMARY:
This is an open label study lung nodules that are either cancer or non-cancer and who are eligible for surgical resection. Patients will undergo their surgery with the help of the Lung Resection Marker Locator Kit which will assist the surgeon in both the location and resection of the lung nodule under real-time guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 21 years or older as it is extremely rare for younger people to be at risk for lung cancers.
2. Be deemed candidates for the lung resection surgery, which will be determined by their treating Thoracic Surgeon (also a physician investigator)
3. Have lesions that are nodules/GGO or other abnormal opacity that can be accurately measured in at least one dimension using conventional techniques
4. Seen at BWH Thoracic Surgery outpatient clinics or as inpatient (Note: Subjects will be formally consented to the study at BWH only)

Exclusion Criteria:

1. Female subjects pregnant or breastfeeding
2. Subjects with a pacemaker or equivalent devices (AICD) due to the use of electromagnetic tracking generator.
3. Patients who are not scheduled for lung surgery

   -

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
To compare the measurements from the J-bar fiducial to the first staple line obtained by the device in vivo to that performed in the frozen section room on the lung specimen obtained (which includes both the J bar and the staple line). | 1 day
  device feasibility

SECONDARY OUTCOMES:
whether coefficient is needed | 1 day
  To determine whether a coefficient needs to be defined to harmonize the distance measured with the device to that found by pathologists
time required for device placement | 1 day
  3. To determine the length of time needed for the placement of the device and record measurements.
demonstrate safe surgical remove of lung nodule | 30 day
  no increased surgical morbidity from the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States